CLINICAL TRIAL: NCT07302256
Title: A Randomized, Double-blind, Controlled Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of the Influenza Virus Split Vaccine for Individuals Aged 60 Years and Above
Brief Title: A Clinical Trial of Influenza Virus Split Vaccine for Individuals Aged 60 Years and Above
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIBP-V05-001
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Influenza
Keywords: Influenza virus split vaccine; The elderly; Immunogenicity; Safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (Experimental): Influenza virus split vaccine, with a specification of 0.7mL/bottle
  Interventions: Biological: Influenza virus split vaccine (0.7mL/vial)
- Control group 1 (Active Comparator): Influenza virus split vaccine, with a specification of 0.5mL/bottle
  Interventions: Biological: Influenza virus split vaccine
- Control group 2 (Placebo Comparator): Phosphate buffer solution
  Interventions: Biological: Phosphate buffer solution (PBS)

INTERVENTIONS:
Biological: Influenza virus split vaccine (0.7mL/vial) — Influenza virus split vaccine, with a specification of 0.7mL/bottle, containing 60 μ g of hemagglutinin from H1N1, H3N2, and B influenza virus strains each
  Arms: Experimental group
Biological: Influenza virus split vaccine — Influenza virus split vaccine, with a specification of 0.5mL/bottle, containing 15 μ g of hemagglutinin from H1N1, H3N2, and B influenza virus strains each
  Arms: Control group 1
Biological: Phosphate buffer solution (PBS) — PBS, with a specification of 0.5mL/bottle.
  Arms: Control group 2

SUMMARY:
This is a randomized, blinded, controlled phase I clinical trial with a total of 120 participants aged ≥ 60 years. Experimental group: Influenza virus split vaccine (0.7mL/vial), control group 1: Influenza virus split vaccine, control group 2: placebo group. The three groups were recruited at a ratio of 1:1:1, and 40 individuals were randomly vaccinated in each group. Each person was injected with one dose of the vaccine into the deltoid muscle of the upper arm. Participants in each study group are required to undergo laboratory indicator tests before and on the 4th day after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years old, gender not limited, and able to provide legal identification;
* Volunteers voluntarily participate in the study and sign an informed consent form;
* Volunteers have the ability to understand research procedures, use thermometers, scales, and fill out diary cards as required, and can participate in all planned follow-up visits.

Exclusion Criteria:

* On the day of enrollment, the axillary temperature was ≥ 37.3 ℃;
* Those who have had influenza in the past 6 months or meet the definition of influenza like cases;
* Have received any influenza vaccine within the past 12 months or have planned to receive any influenza vaccine during the study period;
* Allergies to any components of the research vaccine, history of allergic reactions to the use of gentamicin sulfate, history of severe allergies to any vaccine/drug, or history of asthma;
* Suffering from a serious illness that prevents the completion of the entire study; Within 3 days prior to vaccination, there is an acute illness or an acute exacerbation of a chronic disease;
* Have used antipyretic or analgesic drugs or anti allergic drugs within 3 days before vaccination;
* Have received any vaccine within 2 weeks prior to vaccination;
* Have received immunosuppressive therapy or other immunomodulatory drugs within 6 months prior to receiving the experimental vaccine, For example, immunosuppressive doses of glucocorticoids, monoclonal antibodies, thymosin, interferon, etc., or planned to receive such treatment within one month after the first dose of vaccination to full immunization, but local medication is allowed;
* Suffering from congenital or acquired immunodeficiency, human immunodeficiency virus (HIV) infection, lymphoma, leukemia, or other autoimmune diseases;
* Suffering from serious chronic diseases, serious cardiovascular diseases, such as hypertension that cannot be controlled by drugs, diabetes that cannot be controlled by drugs or has serious complications, liver and kidney diseases, pulmonary edema, malignant tumors, etc;
* Have received blood or blood related products within the past 6 months;
* Individuals with progressive neurological disorders, including a history of seizures, epilepsy, encephalopathy, Guillain Barr é syndrome, psychiatric or family history;
* Have a history of abnormal coagulation function and have been using anticoagulants within 3 weeks before vaccination;
* Patients with splenectomy, functional splenectomy, splenectomy, or other important organ resection or partial resection;
* Plan to move before the end of the study or leave the local area for a long time during the scheduled study visit;
* Currently or recently planning to participate in other clinical trials;
* Abnormal laboratory test indicators before vaccination;
* Researchers determine any situation that is not suitable for clinical trials.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Unsolicited Adverse Events | 30 days after vaccination
  Other adverse events that occurred among participants within 0-30 days after vaccination, in addition to the solicited adverse events.
Solicited Adverse Events (AEs) | 7 days after vaccination
  Adverse events defined by the protocol that occurred to the participant during 0-7 days after vaccination.
Serious Adverse Events (SAE) | 6 months after vaccination
  That is serious adverse events, any serious adverse events that occurred to the participant during the study period.

SECONDARY OUTCOMES:
Seroconversion rate | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, the HI antibody seroconversion rate against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Ratio of ≥1:40 | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, the ratio of HI antibody titers ≥ 1:40 against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Geometric mean titer (GMT) | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, GMT of HI antibodies against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.
Geometric mean increase (GMI) | 30 days after vaccination
  30 days after vaccination of all participants with the experimental vaccine or control vaccines, GMI of HI antibodies against any subtype of influenza virus in the experimental vaccine group or the control vaccine groups.

CONTACTS AND LOCATIONS:
Overall Officials: Yeqing Tong, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Danjiangkou Disease Prevention and Control Center, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No